CLINICAL TRIAL: NCT03103360
Title: Relationship Between the Pupillary Pain Index Measured One Minute Before Incision and the Motor, Hemodynamic and Electroencephalographic Reaction to Skin Incision in Patients Under General Anesthesia
Brief Title: Pupillary Pain Index and Reaction to Skin Incision
Status: Completed | Type: Observational
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Other Study IDs: PPI incision
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Pain; Anesthesia; Surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: videopupillometer — Measure of pupillary diameter and pupillary pain index via an infrared camera Each measure lasts approximately 20 seconds
Procedure: skin incision — performed under general anesthesia by the surgeon, at the beginning of an elective or emergency surgery.

SUMMARY:
During routine general anesthesia (not standardized, left to the discretion of the attending anesthesiologist), pupillary pain index was measured one minute before skin incision. Then, variations in heart rate, blood pressure and bispectral index during the three minutes following skin incision were recorded, as well as the occurrence of movements.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring general anesthesia
* surgical procedure involving a skin incision
* no regional anesthesia
* written informed consent

Exclusion Criteria:

- neurologic or ophthalmic disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under general anesthesia for an elective or emergent surgery requiring a skin incision in a body area not covered by regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
Relationship between pre-incision pupillary pain index and post-incision heart rate increase | 4 minutes: one minute before incision, 3 minutes after incision
Relationship between pre-incision pupillary pain index and post-incision blood pressure increase | 4 minutes: one minute before incision, 3 minutes after incision
Relationship between pre-incision pupillary pain index and post-incision bispectral index increase | 4 minutes: one minute before incision, 3 minutes after incision
Relationship between pre-incision pupillary pain index and post-incision movement occurrence | 4 minutes: one minute before incision, 3 minutes after incision

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, MD-PHD, Study Director — University Hospital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No